CLINICAL TRIAL: NCT05997706
Title: Unraveling the Klinefelter's Disease Physiopathology by Organoid Model
Brief Title: Unraveling the Klinefelter's Disease Physiopathology
Acronym: KLINEFELTER
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2018/27AVR/196
Record Dates: First submitted 2019-06-27; First posted 2023-08-18 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: Klinefelter Syndrome; Infertility, Male
Keywords: Klinefelter Syndrome; fertility preservation, male
MeSH Terms: conditions — Klinefelter Syndrome; Infertility, Male

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Infertile patients (Experimental): Infertile patients going to surgery for fertility preservation or infertility treatment at University Clinic Saint-Luc Brussels
  Interventions: Procedure: Testicular biopsy

INTERVENTIONS:
Procedure: Testicular biopsy — Testicular biopsy is a clinical procedure for extraction of testicular tissue

SUMMARY:
Organoid Model to unravel Klinefelter Syndrome infertility

Klinefelter Syndrome (KS) is characterized by the presence of an extra chromosome X in male (47,XXY), it is the most frequent genetic cause of azoospermia in adult men. The investigators will isolate and expand spermatogonial cells from KS patients, then using an organoid model investigators will compare the behavior of these Spermatogonia from KS patients when interacting with four combinations of somatic cell types incorporated in the Extra Cellular Matrix hydrogel.

DETAILED DESCRIPTION:
Men with Klinefelter Syndrome candidate for TESE or microTESE (testicular sperm extraction) for azoospermia.

One extra testicular biopsy (1-2 mm) will be cryopreserved and used later for the cells isolation and culture.

ELIGIBILITY:
Inclusion Criteria:

* Klinefelter

Exclusion Criteria:

* Mosaicism

Ages: 5 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 20 (Estimated)
Dates: Start 2018-06-12 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Klinefelter's infertility physiopathology | Up to 60 days with intermediate time analyses at the 5th and 10 th passage of cultures.
  Testicular biopsies will be digested using two steps enzymatic protocol. Cell suspensions will be in vitro cultured during 2 months. The following analyses will be performed: cells counts, cells characterisation by immunofluorescence and RTqPCR specific for the cell type, cells karyotypes.

CONTACTS AND LOCATIONS:
Overall Officials: Christine Wyns, MD, PhD, Principal Investigator — Cliniques Universitaires St Luc
Locations (1):
- Cliniques Universitaires St Luc, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Giudice MG, Kanbar M, Poels J, Duquenne A, Wyns C. Long-term culture of human Sertoli cells from adult Klinefelter patients as a first step to develop new tools for unravelling the testicular physiopathology. Hum Reprod. 2024 Nov 1;39(11):2400-2410. doi: 10.1093/humrep/deae201. PMID 39237101